CLINICAL TRIAL: NCT06129032
Title: Comparing Quadratus Lumborum Type 1 Block to The Combination Of Intraperitoneal Instillation Of Local Anesthetics And Wound Infiltration For Postoperative Pain After Cesarean Delivery: A Prospective Double-Blind Randomized Controlled Study
Brief Title: Comparing QLB Type I Block to Intraperitoneal Instillation Added to Wound Infiltration for Postoperative Cesarian Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Clinical Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/462
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Wound infiltration + Intraperitoneal local anaesthetic instillation (Active Comparator): the surgeon will be given a solution containing 20 ml of 0.5% bupivacaine, 20 ml of 2% lidocaine and 1:200,000 epinephrine with a total volume of 40 ml. A volume of 10 millilitres of the solution will be administered through the drip technique into each of the four quadrants of the uterus prior to the subsequent closure of the parietal peritoneum or fascia. A total volume of 10 ml of the solution will be administered through infiltration at the edges of the rectus aponeurosis, while the remaining 20 ml will be infiltrated subcutaneously into the incision. Patients will receive 800mg of ibuprofen and 1g of paracetamol 30 minutes prior to the end of the procedure. Following the surgical procedure, each patient will get a dosage of 15 mg/kg paracetamol every 6 hours and 800 mg of ibuprofen every 8 hours for 24 hours.
  Interventions: Procedure: Wound infiltration (LWI) + Intraperitoneal local anaesthetic (IPLA) instillation
- Group QUADRATUS LUMBORUM BLOCK (Active Comparator): In the QLB group, quadratus lumborum type 1 block will be applied bilaterally on both sides with a total of 40 ml of solution containing 20 ml of 0.5% bupivacaine + 20 ml of 2% lidocaine + 1:200.000 epinephrine, under ultrasound guidance. Patients will receive 800mg of ibuprofen and 1g of paracetamol 30 minutes prior to the end of the procedure. Following the surgical procedure, each patient will get a dosage of 15 mg/kg paracetamol every 6 hours and 800 mg of ibuprofen every 8 hours for 24 hours.
  Interventions: Procedure: Group QUADRATUS LUMBORUM BLOCK (QLB)

INTERVENTIONS:
Procedure: Wound infiltration (LWI) + Intraperitoneal local anaesthetic (IPLA) instillation — a solution containing 20 ml of 0.5% bupivacaine, 20 ml of 2% lidocaine and 1:200,000 epinephrine with a total volume of 40 ml. A volume of 10 millilitres of the solution will be administered through the drip technique into each of the four quadrants of the uterus prior to the subsequent closure of the parietal peritoneum or fascia.
  A total volume of 10 ml of the solution will be administered through infiltration at the edges of the rectus aponeurosis, while the remaining 20 ml will be infiltrated subcutaneously into the incision
  Arms: Group Wound infiltration + Intraperitoneal local anaesthetic instillation
Procedure: Group QUADRATUS LUMBORUM BLOCK (QLB) — quadratus lumborum type 1 block will be applied bilaterally on both sides with a total of 40 ml of solution containing 20 ml of 0.5% bupivacaine + 20 ml of 2% lidocaine + 1:200.000 epinephrine, under ultrasound guidance
  Arms: Group QUADRATUS LUMBORUM BLOCK

SUMMARY:
This study aimed to compare the efficacy of local anaesthetic infiltration into all layers of the anterior abdominal wall with peritoneal instillation and QLB type I for pain reduction in women undergoing elective cesarean section under spinal anaesthesia.

DETAILED DESCRIPTION:
This study will be conducted as a prospective randomized, controlled, double-blind trial following the approval of the ethical committee at Atatürk University Medical Faculty Hospital and after obtaining written consent from the participating patients. The study will include pregnant women aged 18 to 50 with American Society of Anesthesiologists (ASA) II classification, full-term and singleton pregnancies planned to undergo cesarean section using Pfannenstiel incision with spinal anaesthesia. Using a randomisation procedure, the participants will be allocated into two equal groups: Group IPLA+ LWI and Group QLB.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 to 50
* American Society of Anesthesiologists (ASA) II classification,
* full-term and singleton pregnancies planned to undergo cesarean section
* using Pfannenstiel incision
* spinal anaesthesia

Exclusion Criteria:

* whom neuraxial anaesthesia is contraindicated,
* those who are allergic to drugs to be used in the study,
* who refused to participate in the study,
* those with BMI>35 kg/m2,
* ASA score ≥3 or higher,
* diabetes mellitus, preeclampsia, cardiovascular disease, chronic pain and neuropathic pain,
* individuals who have received opioids during the surgical procedure for intraoperative pain,
* patients who have undergone abdominal surgery,
* patients who have experienced a transition from spinal anaesthesia to general anaesthesia due to failure,
* those with excessive bleeding during the operation,
* who have uterine atony,
* those who have a drain placed in the area to be infiltrated,
* those who cannot understand the Visual Analog Scale (VAS),
* who have a history of drug addiction and psychiatric disorder

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
difference between total opioid consumption in 24 hours | postoperative 24 hours
  The study will involve monitoring the intake of opioids at specific time intervals (2nd, 4th, 6th, 12th, and 24th hours), calculating the cumulative opioid consumption until the 24th hour

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Dostbil, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Bateman BT, Franklin JM, Bykov K, Avorn J, Shrank WH, Brennan TA, Landon JE, Rathmell JP, Huybrechts KF, Fischer MA, Choudhry NK. Persistent opioid use following cesarean delivery: patterns and predictors among opioid-naive women. Am J Obstet Gynecol. 2016 Sep;215(3):353.e1-353.e18. doi: 10.1016/j.ajog.2016.03.016. Epub 2016 Mar 17. PMID 26996986
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500